CLINICAL TRIAL: NCT06436508
Title: The Investigation of the Impact of Early Mobilization on the Outcome, the Appearance of Early Ischemic Damage, the Functional Status, and the Length of Intensive Care Treatment in Patients With Aneurysmal Subarachnoid Hemorrhage.
Brief Title: The Investigation of the Impact of Early Mobilization on the Outcome in Patients With Aneurysmal Subarachnoid Hemorrhage.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Collaborators: National Institute of Mental, Neurological and Neurosurgery (Unknown); Borsod-Abaúj-Zemplén County Central Hospital and University Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, Péter Csécsei, Assistant Professor, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HunSAHEMob
Record Dates: First submitted 2024-02-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Early Ambulation; Standard of Care; Subarachnoid Hemorrhage, Aneurysmal
Keywords: subarachnoid hemorrhage; early mobilization
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization (Experimental): This group is mobilized in the intensive care unit by the institutional physiotherapist with the assistance of specialized personnel. Mobilization is carried out according to the Early Mobilization Protocol (EMP)
  Early mobilization protocol:
  * Step 1 - Day 1: Bed rest, elevation of the head end to 30°
  * Step 2 - Day 2: Bed rest, elevation of the head end to 60°
  * Step 3 - Day 3: Bed rest, elevation of the head end to 80°
  * Step 4 - Day 4: Sitting on the edge of the bed
  * Step 5 - Day 5: Sitting in a chair, standing up
  * Step 6 - Day 6: Walking with or without assistance
  * Step 7 - Day 7: Walking with or without assistance from today
  Interventions: Behavioral: Early mobilization protocol
- Standard bed rest (Active Comparator): No early mobilization
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Early mobilization protocol — * Step 1 - Day 1: Bed rest, elevation of the head end to 30°
  * Step 2 - Day 2: Bed rest, elevation of the head end to 60°
  * Step 3 - Day 3: Bed rest, elevation of the head end to 80°
  * Step 4 - Day 4: Sitting on the edge of the bed
  * Step 5 - Day 5: Sitting in a chair, standing up
  * Step 6 - Day 6: Walking with or without assistance
  * Step 7 - Day 7: Walking with or without assistance from today
  Arms: Early mobilization
Behavioral: Standard care — During standard care, early mobilization does not take place in the intensive care unit; the patient receives only standard supportive care in bed rest.
  Arms: Standard bed rest

SUMMARY:
The goal of the randomized clinical trial is to examine the effect of early mobilization on primary and secondary outcomes in patients with subarachnoid hemorrhage caused by aneurysm rupture.

Researchers will compare early mobiliziation vs. standrad bed rest care.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 ys
* Premorbid modified Rankin Scale score of 0-2
* WFNS I-IV at enrollment
* Aneurysm occlusion has occurred through open or endovascular means
* Minimum 24 hours elapsed after aneurysm occlusion
* The patient has not received thrombolytic therapy
* Vital parameters are appropriate (mean arterial pressure [MAP] >80 or >110 mm Hg)
* Signed patient information and consent form
* Enrollment occurs within 72 hours following ictus

Exclusion Criteria:

* Age under 18 years
* Traumatic subarachnoid hemorrhage
* Incapacitated or limited capacity for action before ictus
* Confirmed pregnancy
* Aneurysm multiplicity (unless all aneurysms are treated)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Disability in early mobilization group (EM) vs. standard care group (SC) - modified Rankin score | 14 day; 3 months
  Outcome assessments will include:
  Modified Rankin Scale
  Disability is assessed by the modified Rankin Scale, dichotomized at a score of 0 to 3 versus 4 to 6 (6=death).Assessment is performed by a blinded investigator of the local study center by personal visit.
Disability in early mobilization group (EM) vs. standard care group (SC) - Extended Glasgow Outcome Scale | 14 day; 3 months
  Extended Glasgow Outcome Scale
  Description of the neurological outcome by using extended Glasgow Outcome Score
  1. Death
  2. Vegetative sate
  3. Lower severe disability
  4. Upper severe disability
  5. Lower moderate disability
  6. Upper moderate disability
  7. Lower good recovery
  8. Upper good recovery
  Assessment is performed by a blinded investigator of the local study center by personal visit.

SECONDARY OUTCOMES:
Onset of delayed cerebral ischemia (DCI) | 3-21 days
  Occurence of DCI after aneurysmal subarachnoid hemorrhage
Onset of severity of macrovascular vasospasm | Up to 14 days
  based on cerebral vasospasm grade
  Grade 0 All intracranial vessels show a physiological shape Grade 1 Vasospasm affects the A2, A1, and M2 segments Grade 2 Vasospasm expands to the M1 and terminal segment of the internal carotid artery Grade 3 Severe reduction in the intradural internal carotid artery with filiform A1 and M1 segments, which sometimes appears like a ghost (ghost sign)
Stay in the Intensive Care Unit (ICU) | Up to 28 days
  Length of stay in the Intensive Care Unit (ICU)
Type of post-hospital discharge placement | Up to 30 days
  home discharge, rehabilitation, chronic care, etc.
Readmission to the ICU | Up to 30 days
  repeated ICU treatment following ward discharge
Occurrence of infection and its time in the intensive care unit | Up to 30 days
  infection and its time in the intensive care unit
Barthel score | 14 day; 3 months
  For assessing activities of daily living in patients with aneurysmal subarachnoid hemorrhage; ordinal scale rates bowel function, bladder function, grooming, toilet use, feeding independence, transfer independence, mobility, dressing ability, stair use, and bathing ability to tabulate a composite score ranging from 0 to 100. Score of 100 represents totally independent.
  Assessment is performed by a blinded investigator of the local study center by personal visit.
Functional Independence Measure (FIM) scale | 14 day
  The FIM's assessment of degree of disability depends on the patient's score in 18 categories, focusing on motor and cognitive function. Each category or item is rated on a 7-point scale (1 = <25% independence; total assistance required, 7 = 100% independence)
  Assessment is performed by a blinded investigator of the local study center by personal visit.
Montreal Cognitive Assessment (MoCA) | 14 day; 3 months
  MoCA scores range between 0 and 30.
  The MoCA is used for assessment for detecting cognitive impairment. A score of 26 or over is considered to be normal.
  Assessment is performed by a blinded investigator of the local study center by personal visit.
Hospital Anxiety and Depression Scale (HADS) | 14 day; 3 months
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.
  Assessment is performed by a blinded investigator of the local study center by personal visit.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Csecsei, MD. PhD, Principal Investigator — University of Pecs
Locations (3):
- Hungary (3):
  - University of Pecs, Pécs, Baranya
  - Central Hospital of B.A.Z. County, Miskolc, BAZ
  - National Institute of Mental Health, Neurology, and Neurosurgery, Budapest

IPD SHARING:
Plan to Share IPD: Yes
Investigators will use external resources for an appropriate repository for their data
Supporting Information: Study Protocol, SAP
Time Frame: After study completion for 3 years.
Access Criteria: upon reasonable request